CLINICAL TRIAL: NCT02878655
Title: Evaluation of the Overall Quality of Life After the Neck Dissection Retro-spinal Sector (IIb), in Squamous Cell Carcinomas Clinical and Radiological N0 VADS
Acronym: QDV2b
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 14-059
Record Dates: First submitted 2016-05-27; First posted 2016-08-25 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: SCCHN
Keywords: N0 clinical and radiological; dissection IIb sector

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The nodal involvement in squamous cell carcinomas of the upper aerodigestive tract (VADS) is one of the main factors of poor prognosis, justifying the surgical management of neck dissection as a reference treatment.

Under the influence of the American Hayes Martin, it was considered until the 1960s that "over the intervention was, the greater the chance of recovery was". But has since been developed by the Argentine Osvaldo Suarez the concept of functional course, which consists of resection of lymph node tissue while retaining the main structures (muscles, nerves, vessels), as opposed to the recess radical which is reserved for the invasive metastasis.

In addition to these notions, our job is to evaluate the quality of life of patients with SCCHN, N0 clinical and radiological, enjoying a functional neck dissection including IIb sector to support the approach which would be to stop the systematic inclusion of this territory.

ELIGIBILITY:
Inclusion Criteria:

* Patient with SCCHN histologically proven N0 clinical and radiological
* Neoplastic Location: oral cavity, oropharynx, hypopharynx, larynx
* Patient candidate for a neck dissection fonctonnel
* Life expectancy> 3 months
* Stable patient not exhibiting at the time of recurrence sign of examination or other scalable neoplasia
* Age over 18 ans
* Patient was informed of the study
* Patient fluent French

Exclusion Criteria:

* Patients with a history of malignancy, outside a basal cell cancer or cancer of the neck treated and cured
* Patient has at the time of examination of recurrence of signs or other scalable neoplasia
* Uncontrolled Infectious diseases
* Neoadjuvant radiotherapy
* Patient nursing or pregnant or lack of contraception during their reproductive
* Intercurrent pathology involving life-threatening
* Any medical or psychological condition associated that could compromise the patient's ability to participate in the study
* Inability to submit to medical follow-up study for geographical, social or psychic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SCCHN, N0 clinical and radiological, enjoying a dissection IIb sector
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Visual Annalogue Scale for Global Quality of Life | change over baseline and month 6
  (rate between 0 and 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France